CLINICAL TRIAL: NCT02069340
Title: POPULATION PHARMACOMETRICS FOR ASSESSING RISK OF BISPHOSPHONATE-RELATED OSTEONECROSIS OF THE JAW (BRONJ)
Brief Title: Genetics in Predicting Risk of Bisphosphonate-Related Osteonecrosis of the Jaw in Patients With Cancer Receiving Zoledronic Acid
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 0S-13-3; NCI-2014-00207 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 0S-13-3 (Other: USC Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2014-02-07; First posted 2014-02-24 (Estimated); Last update posted 2017-04-11 (Actual); Status verified 2017-04

CONDITIONS: Malignant Neoplasm; Musculoskeletal Complications
MeSH Terms: conditions — Neoplasms | interventions — Zoledronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (zoledronic acid over 15 minutes) (Experimental): Patients receive zoledronic acid IV over 15 minutes on day 1.
  Interventions: Drug: zoledronic acid; Other: pharmacological study
- Arm II (zoledronic acid over 30 minutes) (Experimental): Patients receive zoledronic acid IV over 30 minutes on day 1.
  Interventions: Drug: zoledronic acid; Other: pharmacological study

INTERVENTIONS:
Drug: zoledronic acid — Given IV
  Other Names: CGP 42446; CGP42446A; NDC-zoledronate; zoledronate; Zometa
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
This randomized clinical trial studies genetics in predicting risk of bisphosphonate-related osteonecrosis of the jaw in patients with cancer receiving zoledronic acid. Zoledronic acid is an anti-resorptive drug used as part of cancer treatment. A serious side effect of these drugs is death of the jawbone, commonly called bisphosphonate-related osteonecrosis of the jaw (BRONJ). Genetic research may help doctors understand risk factors for BRONJ or who is more likely to get BRONJ and why.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To develop a pharmacometric model to predict jawbone zoledronic acid (Zol) concentrations in oncologic patients by conducting a prospective cohort study of Zol pharmacometrics in BRONJ patients, measuring drug in plasma, urine, and jawbone tissue obtained during surgical treatment for BRONJ.

SECONDARY OBJECTIVES:

I. To clinically assess and validate our predictive pharmacometric model, and develop a risk model for BRONJ in oncologic patients receiving intravenous Zol.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive zoledronic acid intravenously (IV) over 15 minutes on day 1.

ARM II: Patients receive zoledronic acid IV over 30 minutes on day 1.

After completion of study treatment, patients are followed up for 1 month.

ELIGIBILITY:
Inclusion Criteria:

* PATIENTS WITH BRONJ:
* All cancer patients > 18 years of any ethnicity who have been treated with intravenous zoledronate (zoledronic acid) for >=1 year duration
* Clinical diagnosis of BRONJ subsequent to oral surgery as established by standard clinical protocol per American Association of Oral and Maxillofacial Surgeons (AAOMS) diagnostic criteria
* Willingness to have photographs taken to document lesions
* Consent for sample collection for urine, hematology, histopathology and microbial profiling
* Cognitively able and willing to provide consent
* Have a World Health Organization (WHO)/Eastern Cooperative Oncology Group (ECOG) performance score =< 2 and life expectancy > 6 months
* PATIENTS WITHOUT BRONJ:
* Cancer patients without BRONJ who have been treated with intravenous zoledronate for >= 1 year duration
* No signs or symptoms of BRONJ
* Willingness to provide consent for sample collection for blood, urine and saliva

Exclusion Criteria:

* WHO/ECOG performance score > 2 and life expectancy of < 6 months
* Coagulopathy
* Active systemic infection or autoimmune disease
* Currently pregnant or within 3 months post-partum, or unwilling to undergo pregnancy testing or report possible pregnancy promptly
* Severe cardiovascular, pulmonary or other systemic conditions that prevent participation in the study
* Salivary gland hypofunction regardless of underlying pathology
* Neutropenia (serum absolute neutrophil count [ANC] < 1,000/uL)
* Cognitive, language or hearing problems
* Renal disease, and we will use a calculated serum creatinine clearance over 30 ml/min at the screening appointment as an exclusion criteria
* Participation in another research project that might interfere with completion of this study
* Patients undergoing active antibiotic therapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-06 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Plasma concentrations of Zol collected at visits 2, 3, 4, and 5 | Up to 1 month
  Data will be iteratively fit to the model using non-parametric modeling, simulation, and clinical dosing software. The parameters will be estimated, as well as their relationships to each other. Each measured patient concentration is Fisher weighted.
Urine concentrations of Zol collected at visits 2, 3, 4, and 5 | Up to 1 month
  Data will be iteratively fit to the model using non-parametric modeling, simulation, and clinical dosing software. The parameters will be estimated, as well as their relationships to each other. Each measured patient concentration is Fisher weighted.
Jawbone tissue concentrations of Zol collected during surgical treatment for BRONJ | Up to 1 month
  Data will be iteratively fit to the model using non-parametric modeling, simulation, and clinical dosing software. The parameters will be estimated, as well as their relationships to each other. Each measured patient concentration is Fisher weighted.

SECONDARY OUTCOMES:
Identify potential risk factors for BRONJ | Up to1 month
  The magnitude of associations between the study variables and BRONJ status will be estimated. For categorical variables, the univariate association with each variable and with BRONJ will be determined using Wald's test of association. For continuous variables, the association with each variable and BRONJ will be determined using Wald's test. Logistic regression will be used to evaluate the risk of BRONJ for development of the final risk model.

CONTACTS AND LOCATIONS:
Overall Officials: Parish Sedghizadeh, Principal Investigator — University of Southern California
Locations (2):
- United States (2):
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - J.Craig Venter Institute-San Diego, San Diego, California